CLINICAL TRIAL: NCT05125419
Title: Serum Homocysteine Level in the Setting of Acute Coronary Syndrome in Young Adult Patients
Brief Title: Homocysteine in Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelnasser Labib, Principal investigator, Sohag University
Other Study IDs: Homocysteine level
Record Dates: First submitted 2021-11-06; First posted 2021-11-18 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Homocysteine level — diagnostic test
  Other Names: HCY

SUMMARY:
This study aims to determine the relation between high homocysteine levels and increased incidence of acute coronary syndrome in young patients

DETAILED DESCRIPTION:
Cross sectional study to:

assess homocysteine level in young adult patients presenting with acute coronary syndrome

ELIGIBILITY:
Inclusion Criteria:

1. - The patients who presented in the hospital with chest pain consistent with acute coronary syndrome with any of the following features:

   1. Electrocardiogram (ECG) changes:

      * ST elevation
      * ST depression
      * T wave inversion
      * recent left bundle branch block
   2. Troponin T elevation (Norma value < 0.06)

      2- Age: -Between 18- 40 years (Group A) - Age > 40 years (Group B)

      Exclusion Criteria:
      1. Chest pain not consistent with acute coronary syndrome
      2. Chronic kidney disease (CKD)
      3. Rheumatic heart disease (RHD)
      4. Congenital heart disease
      5. Anemia
      6. Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presented with acute coronary syndrome admitted to coronary care unit of Sohag University hospital according to inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Coronary care unit admission with acute coronary syndrome | From date of randomization up to 1 month
  Acute coronary syndrome hospitalization and cardiovascular deathes and estimated hazard ratios (HR) by use of multivariable Cox regression models

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed E Amin, Lecturer, Study Chair — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu J, Quan J, Li Y, Wu Y, Yang L. Blood homocysteine levels could predict major adverse cardiac events in patients with acute coronary syndrome: A STROBE-compliant observational study. Medicine (Baltimore). 2018 Oct;97(40):e12626. doi: 10.1097/MD.0000000000012626. PMID 30290636